CLINICAL TRIAL: NCT03621566
Title: Belgian Central Sleep Apnea REgistry (B-CARE)
Brief Title: Belgian Central Sleep Apnea REgistry
Acronym: B-CARE
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: B322201835950
Record Dates: First submitted 2018-07-05; First posted 2018-08-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Central Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Central Sleep Apnea: Subjects with an apnea/hypopnea index ≥ 15/h of sleep and proportion of non-obstructive events > 50%, derived from polysomnography (diagnostic or during positive airway pressure treatment)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Routine care (registry)

SUMMARY:
This study evaluates different factors that determine the treatment choice and treatment compliance in patients with central sleep apnea. All patients will receive routine care (registry).

DETAILED DESCRIPTION:
Central sleep apnea (CSA) is characterized by intermittent cessation or decrease of airflow and effort of breathing during sleep. The diagnostic criteria for CSA varies according to the type of CSA (e.g. CSA due to cardiac failure, due to a medication, ...).

CSA is defined as: (1) an apnea/hypopnea index ≥ 15 per hour of sleep and (2) the number of central apneas and/or hypopneas is > 50% of the total number of apneas and hypopneas.

Presence of CSA is associated with excessive daytime sleepiness and poor sleep quality. Furthermore, in patients with heart failure, presence of CSA was found to be related to mortality. As yet, however, there is insufficient knowledge on the clinical features, pathophysiological background and consecutive algorithms for treatment. Currently, it is not fully clear whether CSA or the treatment of CSA is related to disease progress.

The aim of this trial is to evaluate the current treatment choices for CSA in Belgium and compliance with and effects of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* An apnea/hypopnea index ≥ 15/h of sleep and proportion of non-obstructive events > 50%, derived from polysomnography (diagnostic or during (PAP) treatment)
* Written informed consent provided

Exclusion Criteria:

- Patients with mental disability making it impossible to understand the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with an apnea/hypopnea index ≥ 15/h of sleep and proportion of non-obstructive events > 50%, derived from polysomnography (diagnostic or during positive airway pressure treatment)
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2028-06-25 (Estimated); Study Completion 2028-06-25 (Estimated)

PRIMARY OUTCOMES:
Treatment choice | 5 years
  Proportion of patients treated with the different treatment modalities

SECONDARY OUTCOMES:
Factors determining treatment choice | 5 years
  Relation between patient and CSA characteristics and the treatment choice
Treatment compliance | 5 years
  Compliance to the different treatment modalities
Short Form 36 Health Survey | 5 years
  To measure eight domains of health
  Content:
  * physical functioning
  * role limitations due to physical health
  * bodily pain
  * general health perceptions
  * vitality
  * social functioning
  * role limitations due to emotional problems
  * mental health
  Number of items: 36 items are included in scoring
  Score interpretation: each item scored on a 0 to 100 range so that the lower and highest possible scores are set at 0 and 100. Scores represent the percentage of total possible score achieved.
Pitssburgh Sleep Quality index | 5 years
  To measure sleep quality and disturbances. Score range: 0-21 points, with lower scores indicating better sleep quality.
Mortality | 5 years
  Proportion of subjects alive with different treatment modalities

CONTACTS AND LOCATIONS:
Overall Officials: Dries Testelmans, MD, PhD, Principal Investigator — UZ Leuven
Locations (14):
- Belgium (14):
  - OLV Ziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
  - UZA, Antwerp
  - AZ Sint-Jan, Bruges
  - CHU Saint-Pierre, Brussels
  - Ghent University Hospital, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - CH Jolimont, La Louvière
  - UZ Leuven, Leuven
  - CHR de la Citadelle, Liège
  - CHU UCL Namur, Namur
  - AZ Glorieux, Ronse
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No